CLINICAL TRIAL: NCT04516356
Title: The Effects of Korean Hand Acupressure on Postoperative Nausea-Vomiting and Retching After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevgi Gür (Other)
Responsible Party: Sponsor-Investigator, Sevgi Gür, Lecturer, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13022260-302.14.05-E.158047
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative nausea and vomiting; Nursing; Acupressure; Thyroidectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study to determine the effect of Korean hand acupressure applied after thyroidectomy on postoperative nausea-vomiting and retching.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Korean hand acupressure will be applied to the experimental group 30 minutes before the induction of anesthesia. After determining the pressure / therapy points associated with nausea and vomiting on the patient's hand, a massage will be made for 3-5 minutes with a diagnostic stick. The seeds will then be fixed at these points with a paper patch. Seeds will not be removed for 24 hours. It will be massaged for 3-5 minutes by pressing the seeds every 3-4 hours and making a curling motion at the same time. At the end of the 24th hour, the application will be terminated.
  Interventions: Other: Korean hand acupressure
- Control Arm (No Intervention): In the control group, no application will be made during and after the surgical intervention, and routine treatment and care will be applied.

INTERVENTIONS:
Other: Korean hand acupressure — According to the working principle of Korean hand acupressure; There are active points and areas in the hands and feet that fit the whole body. The active points on the hands and feet are properly matched to reflect the anatomy of the whole organism. Areas in the body and systems suitable for them are in constant contact. In the patient, the signal wave moves from the damaged point or area and reaches the appropriate point immediately. Thus, changes such as severe pain, skin discoloration, hardening, thickening and thinning in some parts of the skin occur at that point. With the stimulation of the effective point, a treatment wave occurs that heals the sick organ.
  Arms: Intervention Arm

SUMMARY:
The study was planned as a randomized controlled experimental study to determine the effect of Korean hand acupressure applied after thyroidectomy on postoperative nausea-vomiting and retching. After ethics committee approval and institutional permission, 42 patients who applied to the general surgery clinic for thyroidectomy between February 1, 2021 and June 1, 2022 and met the inclusion criteria were included in the study. In the light of academic studies reported within the scope of the planned study, the sample size was determined with the effect size d = 0.942 (effect size), α = 0.05 ( margin of error), 1-β = 0.90 (Power) and G-power package program. It was decided to recruit 42 people (21 people per group). The block randomization method was used to determine the experimental and control groups. Randomization was done by a biostatistician other than the researcher. Patients who met the inclusion criteria and agreed to participate in the study were assigned to the experimental and control groups according to the randomization list. Before the operation, the patient was visited and informed about the purpose, content and the intervention to be applied. After obtaining verbal and written consent from the patients who agreed to participate in the study, the "Individual Characteristics Form" was filled. The first part of the "Patient Follow-up Form" was filled in the experimental and control groups on the day of surgery. Korean hand acupressure was applied to the experimental group 30 minutes before the induction of anesthesia. After determining the pressure/treatment points on the patient's hand due to nausea and vomiting, a 3-5 minute massage was performed with the diagnostic stick. The seeds were then fixed at these points with a paper patch. The seeds were not removed for 8 hours. Massage was done for 3-5 minutes by pressing the seeds every 2 hours and making a curling motion at the same time. At the end of the 8th hour, the application was terminated. The application was made by Sevgi Gür, a researcher trained in Korean hand acupressure. In the control group, no application will be made during and after the surgical intervention, and routine treatment and care was applied. Pain, severity of nausea and vomiting, number of nausea-vomiting and retching, name, dose, frequency and duration of antiemetic drugs used were determined by the researcher at the 2nd, 6th, 12th and 24th hours after the patients in the experimental and control groups applied to the clinic. It was recorded in the second part of the "form". At the end of the 24th hour, the Rhodes Nausea, Vomiting and Retching Index score was evaluated by the researcher.

DETAILED DESCRIPTION:
The universe of the research; patients scheduled for thyroidectomy between February 1, 2021 and June 1, 2022, in the general surgery clinic where the study will be conducted, constituted patients who met the inclusion criteria and agreed to participate in the study. The study was planned as a randomized controlled experimental study. The block randomization method was used to determine the experimental and control groups. Randomization was done by a biostatistician other than the researcher. Patients who met the inclusion criteria and agreed to participate in the study were assigned to the experimental and control groups according to the randomization list. Research data were collected in the general surgery ward of a hospital from February 1, 2021 to June 1, 2022. The independent variable of the research is Korean hand acupressure. The dependent variables of the study were postoperative nausea-vomiting and retching (number and severity), pain severity (Visual Analog Scale-VAS), Rhodes nausea-vomiting and retching index score average. In the study, "Individual Characteristics Form" and "Patient Follow-up Form" prepared by the researcher in line with the literature were used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* According to the American Association of Anesthesiologists (ASA) classification; ASA score I and II,
* Elective surgery,
* Individuals with 2 or more risk factors out of 5 risk factors determined in Koivuranta PONV risk factors
* Patients who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Emergency surgery,
* Using antiemetic, steroid or opioid 24 hours before surgery,
* Not agreeing to participate in the research
* Change in consciousness / acute confusion after surgical intervention,
* Has a mental or psychiatric illness that prevents communication,
* Patients whose post-operative condition is unstable will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain severity | Reported pain severity in the first 24 hours after surgery
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst pain
Postoperative nausea and vomiting severity | Reported nausea and vomiting severity in the first 24 hours after surgery
  Nausea and vomiting severity with Visual Assessment Scale (VAS) Score: 0-10; 0- None, 10- Agonizing
The number of postoperative nausea, vomiting and retching | Reported the number of nausea, vomiting and retching in the first 24 hours after surgery
  The number of nausea, vomiting and retching
Use of antiemetics | In the first 24 hours after surgery
  The name, dose, frequency and time of the antiemetic drugs
Rhodes Nausea Vomiting and Retching Index score | At the end of the 24th hour after surgery
  Evaluation of Rhodes Nausea Vomiting and Retching Index score In order to score the scale, responses to items 1, 3, 6 and 7 are calculated in reverse order; For each answer, they are scored as 0: minimum, 4: most discomfort, and the score obtained from 8 items is added. It is expressed as 32 points, the highest possible value.

SECONDARY OUTCOMES:
Postoperative complications | End of surgery to hospital discharge 5-7 days
  Evaluation of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: İlhan Öztekin, Prof, Principal Investigator — Yeditepe University; Deniz S. Öztekin, Prof, Study Director — Istanbul University - Cerrahpasa; Sevgi Gür, MSC, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Provincial Health Directorate Prof. Dr. Cemil Taşcioğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No